CLINICAL TRIAL: NCT01730989
Title: Controlled Clinical Study on the Activity of the Combination of Isoflavones, Agnocastus and Magnolia Extract in Menopause
Brief Title: Estromineral Serena Plus and Symptomatic Menopause
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rottapharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESP-CPR-0312
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Menopause
Keywords: menopause; Kupperman; hot flushes; isoflavones; magnolia; chaste tree
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estromineral Serena Plus (Experimental): Estromineral Serena Plus is an association of soy isoflavones, Lactobacillus sporogenes, magnolia, chaste tree, Vitamin D3, calcium and magnesium.
  1 tablet oad for 12 weeks
  Interventions: Dietary Supplement: Estromineral Serena Plus
- Estromineral (Active Comparator): Estromineral is an association of soy isoflavones, Lactobacillus sporogenes, Vitamin D3, and calcium.
  1 tablet oad for 12 weeks
  Interventions: Dietary Supplement: Estromineral

INTERVENTIONS:
Dietary Supplement: Estromineral Serena Plus
  Arms: Estromineral Serena Plus
Dietary Supplement: Estromineral
  Arms: Estromineral

SUMMARY:
Oestrogen hormone deficiency in menopause leads to symptoms of which hot flushes, night sweats, insomnia and mood changes are the most frequent and, ultimately, worsen the quality of life. The gradual decline of oestrogen from peri-menopause results in altered function of many neurotransmitters, such as dopamine, melatonin and neuropeptides including beta-endorphins, which modulate the function of the hypothalamus and are involved in body thermoregulation.

In post-menopause, dopaminergic activity is significantly reduced and stimulus of the D2 receptors is effective in relieving hot flushes and in reducing the accompanying psychological symptoms.

The use of hormone replacement therapy, which is generally prescribed in the case of moderate or severe symptoms, is limited due to real contraindications or simply the woman's refusal to take the therapy, despite the presence of symptoms requiring its use.

A food supplement, named Estromineral (E), based on natural ingredients such as isoflavones, the absorption of which is increased by the presence of Lactobacillus sporogenes, and Vitamin D3 and calcium, strengthening bone mineralization, has been found to be effective at reducing vasomotor symptoms.

To potentiate the effect of E on the most frequent symptoms in menopause, it was considered rational to add the extracts of magnolia, active on psycho-affective symptoms, and chaste tree, acting on both hot flushes and psychological symptoms and a new food supplement was developed: Estromineral Serena Plus (ESP).

Estromineral Serena Plus is an association of isoflavones with added Lactobacillus, chaste tree and magnolia, active on menopausal vasomotor symptoms and on psycho-affective symptoms.

ELIGIBILITY:
Inclusion Criteria:

* female menopausal age
* more than 5 hot flushes/day
* mood or sleep changes

Exclusion Criteria:

* hormone replacement therapy

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Kupperman index | up to 12 weeks
  To calculate the Kupperman index, the symptoms were weighted as follows: hot flashes (4), insomnia (2), nervousness (2), and all other symptoms (night sweats, depressed mood (melancholy), dizziness, tiredness, joint and muscular pain, headache, and palpitations (1). The highest potential score is thus 51. The score of hot flashes was based on number of complaints per day: slight (more than 5), moderate (5-10), and severe (more than 10)

SECONDARY OUTCOMES:
Adverse events | 4, 8 and 12 weeks
  Onset duration and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo De Leo, MD, Principal Investigator — Siena University
Locations (1):
- Siena University, Siena, Siena, Italy